CLINICAL TRIAL: NCT00752986
Title: A Randomized,Double-blind,Parallel-group,Multicentre,Phase II Study to Evaluate the Safety and Pharmacological Activity of the Combination of Vandetanib (100 or 300 MG/Daily or Placebo)With Fulvestrant (Loading Dose)in Postmenopausal Advanced BC Patients
Brief Title: ZACtima FASlodex Trial in Postmenopausal Advance Breast Cancer Patients Instead of ZACtima FASlodex Trial
Acronym: ZACFAST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D4200L00009; EUDRACT 2008-000579-12
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
Keywords: ZD6474; Vandetanib; Zactima; Fulvestrant; Faslodex; Breast Cancer; Advanced, Metastatic; Hormone Receptor Positive; Post-Menopausal Patients; post-menopausal women with hormone receptor positive advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — vandetanib; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vandetanib at the dose of 100 mg (Experimental): vandetanib at the dose of 100 mg orally once-daily plus placebo to match vandetanib 300 mg orally once-daily plus fulvestrant LD (500 mg im. at day 1 and 250 mg at day 14, 28 and thereafter every 28th day +/- 3)
  Interventions: Drug: ZD6474 (Vandetanib at the dose of 100 mg); Drug: Fulvestrant; Drug: Placebo to match ZD6474 (Vandetanib at the dose of 300 mg)
- Vandetanib at the dose of 300 mg (Experimental): vandetanib at the dose of 300 mg orally once-daily plus placebo to match vandetanib 100 mg orally once-daily plus fulvestrant LD (500 mg im. at day 1 and 250 mg at day 14, 28 and thereafter every 28th day +/- 3)
  Interventions: Drug: Placebo to match ZD6474 (Vandetanib at the dose of 100 mg); Drug: Fulvestrant; Drug: ZD6474 (Vandetanib at the dose of 300 mg)
- Placebo to match vandetanib 100 mg and 300 mg (Placebo Comparator): placebo to match vandetanib 100 mg orally once-daily plus placebo to match vandetanib 300 mg orally once-daily plus fulvestrant LD (500 mg im. at day 1 and 250 mg at day 14, 28 and thereafter every 28th day +/- 3).
  Interventions: Drug: Placebo to match ZD6474 (Vandetanib at the dose of 100 mg); Drug: Fulvestrant; Drug: Placebo to match ZD6474 (Vandetanib at the dose of 300 mg)

INTERVENTIONS:
Drug: ZD6474 (Vandetanib at the dose of 100 mg) — 100 mg as a once daily oral dose, from Day 1 UNTIL disease progression or unacceptable toxicity or consent withdrawal whichever occurs first
  Other Names: Zactima
  Arms: Vandetanib at the dose of 100 mg
Drug: Placebo to match ZD6474 (Vandetanib at the dose of 100 mg) — Placebo of 300 mg as a once daily oral dose, from Day 1 UNTIL disease progression or unacceptable toxicity or consent withdrawal whichever occurs first
  Arms: Placebo to match vandetanib 100 mg and 300 mg; Vandetanib at the dose of 300 mg
Drug: Fulvestrant — All patients will receive fulvestrant Loading Dose (LD). The Loading Dose regimen is 500mg (2 injections) at day 1, followed by 250mg at day 14, 28 and every 28 days thereafter.
  Other Names: Faslodex
Drug: ZD6474 (Vandetanib at the dose of 300 mg) — 300 mg as a once daily oral dose, from Day 1 UNTIL disease progression or unacceptable toxicity or consent withdrawal whichever occurs first.
  Other Names: Zactima
  Arms: Vandetanib at the dose of 300 mg
Drug: Placebo to match ZD6474 (Vandetanib at the dose of 300 mg) — Placebo of 100 mg as a once daily oral dose, from Day 1 UNTIL disease progression or unacceptable toxicity or consent withdrawal whichever occurs first
  Arms: Placebo to match vandetanib 100 mg and 300 mg; Vandetanib at the dose of 100 mg

SUMMARY:
The primary objective is to assess the event-free survival defined as the time from randomisation to progression, death without progression, loss to follow up, whichever occurred first..

DETAILED DESCRIPTION:
end-point Efficacy: event-free survival (EFS)

ELIGIBILITY:
Inclusion Criteria:

* Post menopausal women with locally advanced or metastatic breast cancer
* Patients may have either measurable or non-measurable disease, as defined by RECIST criteria
* One previous hormone therapy or one previous chemotherapy for advanced disease are allowed (patients who have stable but evident disease after chemotherapy are eligible)
* estrogen receptor positive ER+ and/or progesterone receptor positive PR+ on primary or secondary tumour

Exclusion Criteria:

* Hormone receptor negative tumours (ER and PR negative)
* Presence of life-threatening metastatic visceral disease
* Significant cardiovascular event (e.g. myocardial infarction, superior vena cava [SVC] syndrome, New York Heart Association [NYHA] classification of heart disease ³2) within 3 months before entry, or presence of cardiac disease that in the opinion of
* History of arrhythmia or QTc with Bazett's correction unmeasurable or ≥ 480 msec on screening ECG

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (11):
- Italy (11):
  - Research Site, Avellino
  - Research Site, Benevento
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Monserrato
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Prato
  - Research Site, Roma
  - Research Site, Trento
  - Research Site, Varese

REFERENCES:
- [Background] Ciardiello F, Caputo R, Damiano V, Caputo R, Troiani T, Vitagliano D, Carlomagno F, Veneziani BM, Fontanini G, Bianco AR, Tortora G. Antitumor effects of ZD6474, a small molecule vascular endothelial growth factor receptor tyrosine kinase inhibitor, with additional activity against epidermal growth factor receptor tyrosine kinase. Clin Cancer Res. 2003 Apr;9(4):1546-56. PMID 12684431
- See also: D4200L00009_Clinical_Report_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1442&filename=D4200L00009_CSR_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was prematurely terminated.
Pre-assignment Details: 39 participants were randomized to receive vandetanib or placebo.
Period: Overall Study
Arm/Group | Vandetanib at the Dose of 100 mg | Vandetanib at the Dose of 300 mg | Placebo to Match Vandetanib 100 mg and 300 mg
Started | 16 | 12 | 11
Completed | 11 | 11 | 9
Not Completed | 5 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 2
Not completed — Protocol Violation | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No data were analyzed due to the premature study interruption and sample of patients was too low.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vandetanib at the Dose of 100 mg | Vandetanib at the Dose of 300 mg | Placebo to Match Vandetanib 100 mg and 300 mg | Total
Number analyzed (Participants) | 16 | 12 | 11 | 39
Age, Continuous [Mean (Full Range); unit: years] | 63.6 [44 to 78] | 59.8 [48 to 79] | 59.6 [43 to 74] | 61.3 [43 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 11 | 39
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival
Description: Success rate (patients without progression and still on treatment at 24 weeks
Time Frame: Restaging (RECIST) is carried out at screening and every 3 months during the study until 1 year and than every 6 months until objective disease progression.
Arm/Group | Vandetanib at the Dose of 100 mg | Vandetanib at the Dose of 300 mg | Placebo to Match Vandetanib 100 mg and 300 mg
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Time-To-Progression, Progression-Free Survival, Objective Tumor Response Rate (CR+PR), Disease Control Rate (CR+PR+SD) and Duration of Response (DOR)
Time Frame: as for outcome 1
Arm/Group | Vandetanib at the Dose of 100 mg | Vandetanib at the Dose of 300 mg | Placebo to Match Vandetanib 100 mg and 300 mg
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Overall Survival
Time Frame: Assessments for survival must be made at the 60 day follow-up visit and then every 3 months, unless the patient withdraws consent.
Arm/Group | Vandetanib at the Dose of 100 mg | Vandetanib at the Dose of 300 mg | Placebo to Match Vandetanib 100 mg and 300 mg
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Incidence and Type of Adverse Events (AEs), Clinically Significant Laboratory or Vital Sign Abnormalities and Electrocardiographic (ECG) Changes
Time Frame: Continuous assessment of safety.
Arm/Group | Vandetanib at the Dose of 100 mg | Vandetanib at the Dose of 300 mg | Placebo to Match Vandetanib 100 mg and 300 mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Vandetanib at the Dose of 100 mg | Vandetanib at the Dose of 300 mg | Placebo to Match Vandetanib 100 mg and 300 mg
Serious Adverse Events (participants affected / at risk) | 3/16 | 2/12 | 1/11
Other Adverse Events (participants affected / at risk) | 12/16 | 11/12 | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vandetanib at the Dose of 100 mg (N=16) | Vandetanib at the Dose of 300 mg (N=12) | Placebo to Match Vandetanib 100 mg and 300 mg (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
diabetes complication (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
grade 3 erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
right iliac fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
severe arthralgia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
gastroenteritis. (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
grade 3 diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vandetanib at the Dose of 100 mg (N=16) | Vandetanib at the Dose of 300 mg (N=12) | Placebo to Match Vandetanib 100 mg and 300 mg (N=11)
RIGHT HYPOCHONDRIUM PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
AST ELEVATION (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
RECTAL BLEEDING (General disorders) | 0 (0) | 0 (0) | 1 (1)
HEMORRHOIDS (General disorders) | 0 (0) | 0 (0) | 1 (1)
ANAEMIA (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 1 (1)
HYPERCALCEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTRANSAMINASEMIA (Blood and lymphatic system disorders) | 0 (0) | 2 (5) | 1 (1)
TOOTH ACHE (General disorders) | 0 (0) | 0 (0) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
LEFT EYE PAIN (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 3 (3) | 7 (14) | 0 (0)
MUCOSITIS (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
NAUSEA (General disorders) | 2 (2) | 3 (3) | 0 (0)
VOMITING (General disorders) | 1 (1) | 1 (2) | 0 (0)
HEPATIC TOXICITY (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
INSOMNIA (General disorders) | 0 (0) | 3 (3) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 3 (6) | 6 (11) | 0 (0)
HEADACHE (General disorders) | 1 (1) | 2 (2) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
PIASTRINOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0)
ANOREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 2 (2) | 2 (2) | 0 (0)
HYPERTENSION (Cardiac disorders) | 3 (3) | 2 (4) | 0 (0)
FEVER (General disorders) | 2 (2) | 2 (2) | 0 (0)
ONYCHOPATY (General disorders) | 0 (0) | 1 (1) | 0 (0)
JOINT PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
RIB FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
STOMATITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
NEUROPATHY (ARMS) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (5) | 0 (0)
WEIGHT LOSS (General disorders) | 0 (0) | 1 (1) | 0 (0)
LOSS OF APPETITE (General disorders) | 0 (0) | 1 (1) | 0 (0)
DIZZINESS (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
ANXIOUS-DEPRESSIVE SYNDROME (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
THORACIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
TACHICARDY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
SWEATING (General disorders) | 1 (1) | 0 (0) | 0 (0)
EYE ANGIOEDEMA (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
CYSTITIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
LUMBAR PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
TRANSAMINASE INCREASE (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
PAIN RIGHT THORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
FLUSHING (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
SCALP ERITHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
UMBILICAL MYCOSES (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
HAEMORRHAGIC CYSTITIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERPOTASSEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ARTHRALGIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 1 (2) | 0 (0) | 0 (0)
MUSCOLOSKELETRICAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.